CLINICAL TRIAL: NCT06551909
Title: Radioimmunotherapy in Solid Tumors (Aim 2- Stereotactic Neoadjuvant Radiotherapy for Glioblastoma)
Brief Title: Radioimmunotherapy in Solid Tumors (PNRR-MCNT2-2023-12378239-Aim2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: European Commission (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialità San Giuseppe Moscati (Avellino) (Unknown)
Responsible Party: Principal Investigator, Nadia Di Muzio, Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PNRR-MCNT2-2023-12378239- Aim2
Record Dates: First submitted 2024-08-12; First posted 2024-08-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Neodjuvant Radiotherapy; Ultrahypofractionated Radiotherapy; Stereotactic Radiotherapy (SRT); Simultaneous Integrated Boost (SIB); Image Guidance
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: This is study of feasibility in terms of toxicity of a dose escalation radiotherapy procedure, with 5 patients at each dose level, on 30 patients. The dose will be increased, moving to the next 5 patients, if no more than 1 acute toxicity of grade (G) 4 will be registered.
  The assumption is that the percentage of patients free from cumulative acute toxicity G≥3 (Common Terminology Criteria of Adverse Events-CTCAE- v5.0 scale) at 1 month after the end of treatment should not exceed 30%. A sample size of 30 patients results in a two-sided 95% confidence interval with a width of 0.328 (0.136-0.464) when the sample proportion is 0.300.
  Dropouts will be replaced by patients visited later, so as to reach the expected sample. Serum from 30 healthy volunteers, with sex and age characteristics comparable to the patients, will be collected to compare the level of immune biomarkers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): The 30 patients will receive neoadjuvant stereotactic radiotherapy in 5 fractions delivering 30 GY to PTV and 35-50 GY with Simultaneous Integrated Boost (SIB) to GTV using standard chemotherapy (TMZ) after surgery. GTV will be treated with escalating dose levels from 35 to 50 Gy. Patients will be divided into groups of 5 and will receive in the absence of 2 G4 toxicities per group, the following dose levels: 35-40-42.5-45-47.5 and 50 Gy
  Interventions: Radiation: Neoaddjuvant Stereotactic Radiotherapy with Simultaneous Integrated Boost

INTERVENTIONS:
Radiation: Neoaddjuvant Stereotactic Radiotherapy with Simultaneous Integrated Boost — Patients with Glioblastoma will receive neoadjuvant stereotactic radiotherapy to Planning Target Volume (PTV) to 30 Gy in 5 fractions, and a Simultaneous Integrated Boost delivering 35-50 GY to GTV. Patients will be divided into groups of 5 and will receive (in the absence of 2 G4 toxicities per group), the following dose levels: 35-40-42.5-45-47.5 and 50 Gy. Standard Temozolomide chemotherapy will be prescribed after surgery.
  Other Names: Ultrahypofractionated Radiotherapy

SUMMARY:
This is a prospective multicenter study of hypofractionated radiotherapy for the radiation treatment (RT) of solid tumors and in particular for Glioblastoma (in Aim 2). It is based on the results of ongoing studies at our Institute to validate the efficacy of extremely hypofractionated RT in neoadjuvant settings, which observed immunostimulatory effects of RT and the synergy with immune components. The collaboration between San Raffaele Hospital (Milan), the IRCCS Istituto Nazionale dei Tumori Fondazione G. Pascale (Naples) and the San Giuseppe Moscati Hospital of National Relief and High Specialty (Avellino) will ensure that patient recruitment, treatment and monitoring can be translated into facilities of the National Health System using common procedures. The various departments involved will treat patients with the same methods synergistically exploring the immuno/biological factors related to efficacy (and/or toxicity), based on new radioimmunotherapeutic approaches. Clinical and research activity will be developed jointly, drawing on the expertise in radiotherapy, radiomics, oncology, imaging and immunotherapy skills already available.

DETAILED DESCRIPTION:
This is a prospective multicenter pilot study. Functional and spectroscopic neuroradiological imaging will be adopted for treatment planning. Specialized software will be used to perform radiomic feature extraction and analysis of pre-trained neural networks from the advanced MRI (magnetic resonance imaging) and CT (computed tomography) used for simulation, to identify distribution patterns of aggressive and radioresistant disease areas, with higher probability of disease recurrence, and to intensify the dose on the areas identified as more aggressive, in order to counteract intrinsic radioresistance. The hypofractionated radiotherapy paradigm claims the benefit of reduced treatment times, improved quality of life, better access to specialized treatment centers and potentially improved tumor outcomes with greater disease control and less tumor repopulation. The rationale for neoadjuvant RT is based on the idea of counteracting the tumor's aggressive mechanisms with radiotherapy before the disease is surgically removed, in order to maximize the immunostimulatory potential of RT, and therefore reduce recurrences. Neoadjuvant treatment offers numerous advantages, first of all the ability to adjust the dose to the pathological volume identified by MRI and limit the volume of irradiated healthy brain tissue. Furthermore, the use of imaging derived from functional neuroradiological and spectroscopic techniques for treatment planning would allow us to increase the dose on the areas identified as more aggressive, in order act against intrinsic radioresistance. One of the major risks could be the possibility of developing radionecrosis, but this would not be a cause for concern in the neoadjuvant setting, as all irradiated tissue will then be surgically removed. Patients who agree to participate in the study and who would be candidates for radical surgical treatment, according to the evaluation of the Neurosurgery Department of our Institute, will be treated. These patients will receive neoadjuvant radiation treatment in 5 fractions delivering 30 Gy on PTV and 35-50 Gy on GTV, with a dose-escalation modality that involves increasing the dose to 35-40-42.5-45-47.5-50 Gy in groups of 5 consecutive patients, using standard chemotherapy (TMZ) after surgery.

Current diagnostic brain MRI allows a good definition of the initial disease and its most aggressive areas. Since relapses have always been found to occur in irradiated areas and recent studies have shown that reducing margins does not affect overall survival, smaller margins will be used from GTV to CTV and from CTV to PTV. Therefore, smaller volumes will be generated and treated with hypofractionation. Biological equivalent doses (BED) to the standard prescription will be delivered, with boost to a higher biological equivalent dose, in the most aggressive areas, in order to obtain better local control, maintaining an acceptable level of toxicity and therefore improve the evolution of the disease. CE marked devices (software) will be used according to the approved use, for the definition of the target (CT and MRI) and for the delivery of the treatment (linear accelerators) and the standard drug, which has the authorization for marketing, will be prescribed. Radiomic features related to local response and survival will be identified, to obtain a predictive model. At the same time, we will collect PMBC and patient serum in the biobank to identify presumed immunocorrelated of therapy efficacy and/or predictive biomarkers of response/toxicity to therapy. For comparative purposes, serum from healthy volunteers will also be collected, in numbers equivalent to patients and with sex and age characteristics comparable to the latter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Glioblastoma.
* ECOG performance score 0-2 (defined during the first visit)
* Surgically removable lesion (according to the operability criteria established by the Neurosurgery Unit)

For healthy volunteers, people who are as comparable as possible with the patient population in terms of sex and age will be recruited

Exclusion Criteria:

* Previous stroke
* Presence of another primary and/or metastatic tumor For healthy volunteers also, absence of primary and/or metastatic tumor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | one month
  Incidence of acute toxicity of grade 3 or 4 as maximum toxicity value during the radiation treatment or in any case within a month of the end of SBRT, using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale (toxicity from 0- patients without toxicity to 5-death from toxicity)

SECONDARY OUTCOMES:
Disease Free Survival | From the date of radiotherapy end until the date of first documented clinical progression or date of death from any cause, whichever came first, assessed up to 36 months]
  Absence of disease progression during the follow-up
Cancer Specific Survival | From the date of radiotherapy end until the date of first documented clinical progression or date of death from any cause, whichever came first, assessed up to 36 months]
  Death from disease progression during the follow-up
Overall survival | From the date of radiotherapy end until the date of death from any cause, assessed up to 36 months
  Survival from all causes
Local Relapse Free Survival | From the date of radiotherapy end until the date of local progression or date of death from any cause, whichever came first, assessed up to 36 months
  Local control of the disease (at the treated site)
Intracranial Relapse Free Survival | From the date of radiotherapy end until the date of local progression or date of death from any cause, whichever came first, assessed up to 36 months
  Intracranial control of the disease (glioblastoma recurrence outside the treatment field)
Extracranial Relapse Free Survival | From the date of radiotherapy end until the date of local progression or date of death from any cause, whichever came first, assessed up to 36 months
  Distant metastases
Late toxicity | From three months after the start of radiotherapy until the end of follow-up or death, assessed up to 36 months
  Toxicity developed after three months until the end of follow-up or death, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scale, which displayes grades from 1 to 5, with grade 1 meaning mild toxicity and grade 5 death related to toxicity
Subacute Toxicity | From one up to three months after the start of radiotherapy
  Incidence of acute toxicity of grade 3 or 4 as maximum toxicity value registered from one to three months of the end of SBRT, using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 scale (toxicity from 0- patients without toxicity to 5-death from toxicity)
Incidence of Treatment-Emergent Adverse Events as assessed with brain tumor specific quality of life questionnaires | 36 months
  Survey with the questionnaire of European Organisation for Research and Treatment of Cancer (EORTC) Quality of life of brain tumor patients (EORTC QLQ BN20) which contains 25 questions on patients' quality of life with answers from 1, lowest grade, to 4, highest grade
Incidence of Treatment-Emergent Adverse Events as assessed with functional-social- emotional and general well being questionnaires | 36 months
  Survey with the questionnaire FACT-Br on patients' quality of life with answers from 0, lowest grade, to 4, highest grade
Incidence of Treatment-Emergent Adverse Events as assessed with mental status questionnaires | 36 months
  Survey with the questionnaire Mini Mental Status Examination (MMSE). A score of 24-30 indicates normal abilities, while a lower score indicates cognitive deficit.
Periferic mononuclear blood cells (PMBC) subtypes predictive for disease progression and death | Form the start of radiotherapy up to 6 months
  Identification of immune prognostic factors, studying lymphocyte subpopulations and their impact on the results obtained.

OTHER OUTCOMES:
Radiomics | 36 months
  Evaluation of radiomic characteristics: Mathematical extraction of the spatial distribution of signal intensities and pixel interrelationships of medical images of the patients, to quantify textural information resampled according to International Biomarker Standardization Initiative (IBSI).
Predictive factors for disease progression and death | From radiotherapy end to date of local, regional progression, distant failure, or death, assessed up to 36 months
  To identify potential risk factors, the association of clinical and radiation treatment factors with survival outcomes will be estimated using survival trees, univariate/multivariate Cox regression models

CONTACTS AND LOCATIONS:
Overall Officials: Nadia G Di Muzio, Prof, Principal Investigator — IRCCS San Raffaele Scientific Institute
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study (anonymized individual participant data) are available on request from the corresponding author to researchers who provide a methodologically sound proposal. Requests made to the corresponding author will be evaluated by the Lombardy Territorial Ethics Committee
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: for 2 years after the end of the study
Access Criteria: request from the corresponding author approved by the Lombardy Territorial Ethics Committee

REFERENCES:
- [Result] Thust SC, Heiland S, Falini A, Jager HR, Waldman AD, Sundgren PC, Godi C, Katsaros VK, Ramos A, Bargallo N, Vernooij MW, Yousry T, Bendszus M, Smits M. Glioma imaging in Europe: A survey of 220 centres and recommendations for best clinical practice. Eur Radiol. 2018 Aug;28(8):3306-3317. doi: 10.1007/s00330-018-5314-5. Epub 2018 Mar 13. PMID 29536240
- [Result] Castellano A, Falini A. Progress in neuro-imaging of brain tumors. Curr Opin Oncol. 2016 Nov;28(6):484-493. doi: 10.1097/CCO.0000000000000328. PMID 27649026
- [Result] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Result] Laws ER, Parney IF, Huang W, Anderson F, Morris AM, Asher A, Lillehei KO, Bernstein M, Brem H, Sloan A, Berger MS, Chang S; Glioma Outcomes Investigators. Survival following surgery and prognostic factors for recently diagnosed malignant glioma: data from the Glioma Outcomes Project. J Neurosurg. 2003 Sep;99(3):467-73. doi: 10.3171/jns.2003.99.3.0467. PMID 12959431
- [Result] Brown TJ, Brennan MC, Li M, Church EW, Brandmeir NJ, Rakszawski KL, Patel AS, Rizk EB, Suki D, Sawaya R, Glantz M. Association of the Extent of Resection With Survival in Glioblastoma: A Systematic Review and Meta-analysis. JAMA Oncol. 2016 Nov 1;2(11):1460-1469. doi: 10.1001/jamaoncol.2016.1373. PMID 27310651
- [Result] Lacroix M, Abi-Said D, Fourney DR, Gokaslan ZL, Shi W, DeMonte F, Lang FF, McCutcheon IE, Hassenbusch SJ, Holland E, Hess K, Michael C, Miller D, Sawaya R. A multivariate analysis of 416 patients with glioblastoma multiforme: prognosis, extent of resection, and survival. J Neurosurg. 2001 Aug;95(2):190-8. doi: 10.3171/jns.2001.95.2.0190. PMID 11780887
- [Result] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Result] Brandes AA, Franceschi E, Tosoni A, Blatt V, Pession A, Tallini G, Bertorelle R, Bartolini S, Calbucci F, Andreoli A, Frezza G, Leonardi M, Spagnolli F, Ermani M. MGMT promoter methylation status can predict the incidence and outcome of pseudoprogression after concomitant radiochemotherapy in newly diagnosed glioblastoma patients. J Clin Oncol. 2008 May 1;26(13):2192-7. doi: 10.1200/JCO.2007.14.8163. PMID 18445844
- [Result] Desai K, Hubben A, Ahluwalia M. The Role of Checkpoint Inhibitors in Glioblastoma. Target Oncol. 2019 Aug;14(4):375-394. doi: 10.1007/s11523-019-00655-3. PMID 31290002
- [Result] Gzell C, Back M, Wheeler H, Bailey D, Foote M. Radiotherapy in Glioblastoma: the Past, the Present and the Future. Clin Oncol (R Coll Radiol). 2017 Jan;29(1):15-25. doi: 10.1016/j.clon.2016.09.015. Epub 2016 Oct 13. PMID 27743773
- [Result] Valduvieco I, Verger E, Bruna J, Caral L, Pujol T, Ribalta T, Boget T, Oleaga L, Pineda E, Graus F. Impact of radiotherapy delay on survival in glioblastoma. Clin Transl Oncol. 2013 Apr;15(4):278-82. doi: 10.1007/s12094-012-0916-x. Epub 2012 Jul 24. PMID 22855197
- [Result] Burko P, D'Amico G, Miltykh I, Scalia F, Conway de Macario E, Macario AJL, Giglia G, Cappello F, Caruso Bavisotto C. Molecular Pathways Implicated in Radioresistance of Glioblastoma Multiforme: What Is the Role of Extracellular Vesicles? Int J Mol Sci. 2023 Mar 2;24(5):4883. doi: 10.3390/ijms24054883. PMID 36902314
- [Result] Tang Z, Dokic I, Knoll M, Ciamarone F, Schwager C, Klein C, Cebulla G, Hoffmann DC, Schlegel J, Seidel P, Rutenberg C, Brons S, Herold-Mende C, Wick W, Debus J, Lemke D, Abdollahi A. Radioresistance and Transcriptional Reprograming of Invasive Glioblastoma Cells. Int J Radiat Oncol Biol Phys. 2022 Feb 1;112(2):499-513. doi: 10.1016/j.ijrobp.2021.09.017. Epub 2021 Sep 14. PMID 34534627
- [Result] Pant A, Lim M. CAR-T Therapy in GBM: Current Challenges and Avenues for Improvement. Cancers (Basel). 2023 Feb 16;15(4):1249. doi: 10.3390/cancers15041249. PMID 36831591
- [Result] Weller M, van den Bent M, Preusser M, Le Rhun E, Tonn JC, Minniti G, Bendszus M, Balana C, Chinot O, Dirven L, French P, Hegi ME, Jakola AS, Platten M, Roth P, Ruda R, Short S, Smits M, Taphoorn MJB, von Deimling A, Westphal M, Soffietti R, Reifenberger G, Wick W. EANO guidelines on the diagnosis and treatment of diffuse gliomas of adulthood. Nat Rev Clin Oncol. 2021 Mar;18(3):170-186. doi: 10.1038/s41571-020-00447-z. Epub 2020 Dec 8. PMID 33293629
- [Result] Trone JC, Vallard A, Sotton S, Ben Mrad M, Jmour O, Magne N, Pommier B, Laporte S, Ollier E. Survival after hypofractionation in glioblastoma: a systematic review and meta-analysis. Radiat Oncol. 2020 Jun 8;15(1):145. doi: 10.1186/s13014-020-01584-6. PMID 32513205
- [Result] Lu VM, Kerezoudis P, Brown DA, Burns TC, Quinones-Hinojosa A, Chaichana KL. Hypofractionated versus standard radiation therapy in combination with temozolomide for glioblastoma in the elderly: a meta-analysis. J Neurooncol. 2019 Jun;143(2):177-185. doi: 10.1007/s11060-019-03155-6. Epub 2019 Mar 27. PMID 30919157
- [Result] Liao G, Zhao Z, Yang H, Li X. Efficacy and Safety of Hypofractionated Radiotherapy for the Treatment of Newly Diagnosed Glioblastoma Multiforme: A Systematic Review and Meta-Analysis. Front Oncol. 2019 Oct 14;9:1017. doi: 10.3389/fonc.2019.01017. eCollection 2019. PMID 31681570
- [Result] Kotecha R, Mehta MP. Extreme hypofractionation for newly diagnosed glioblastoma: rationale, dose, techniques, and outcomes. Neuro Oncol. 2020 Aug 17;22(8):1062-1064. doi: 10.1093/neuonc/noaa133. No abstract available. PMID 32479631
- [Result] Azoulay M, Chang SD, Gibbs IC, Hancock SL, Pollom EL, Harsh GR, Adler JR, Harraher C, Li G, Hayden Gephart M, Nagpal S, Thomas RP, Recht LD, Jacobs LR, Modlin LA, Wynne J, Seiger K, Fujimoto D, Usoz M, von Eyben R, Choi CYH, Soltys SG. A phase I/II trial of 5-fraction stereotactic radiosurgery with 5-mm margins with concurrent temozolomide in newly diagnosed glioblastoma: primary outcomes. Neuro Oncol. 2020 Aug 17;22(8):1182-1189. doi: 10.1093/neuonc/noaa019. PMID 32002547
- [Result] Mendoza MG, Azoulay M, Chang SD, Gibbs IC, Hancock SL, Pollom EL, Adler JR, Harraher C, Li G, Gephart MH, Nagpal S, Thomas RP, Recht LD, Jacobs LR, Modlin LA, Wynne J, Seiger K, Fujimoto D, Usoz M, von Eyben R, Choi CYH, Soltys SG. Patterns of Progression in Patients With Newly Diagnosed Glioblastoma Treated With 5-mm Margins in a Phase 1/2 Trial of 5-Fraction Stereotactic Radiosurgery With Concurrent and Adjuvant Temozolomide. Pract Radiat Oncol. 2023 May-Jun;13(3):e239-e245. doi: 10.1016/j.prro.2023.01.008. Epub 2023 Feb 2. PMID 36736621
- [Result] Kumar N, Kumar R, Sharma SC, Mukherjee A, Khandelwal N, Tripathi M, Miriyala R, Oinam AS, Madan R, Yadav BS, Khosla D, Kapoor R. Impact of volume of irradiation on survival and quality of life in glioblastoma: a prospective, phase 2, randomized comparison of RTOG and MDACC protocols. Neurooncol Pract. 2020 Jan;7(1):86-93. doi: 10.1093/nop/npz024. Epub 2019 Jul 18. PMID 32257287
- [Result] Gao X, McDonald JT, Hlatky L, Enderling H. Acute and fractionated irradiation differentially modulate glioma stem cell division kinetics. Cancer Res. 2013 Mar 1;73(5):1481-90. doi: 10.1158/0008-5472.CAN-12-3429. Epub 2012 Dec 26. PMID 23269274
- [Result] Grossman SA, Ye X, Lesser G, Sloan A, Carraway H, Desideri S, Piantadosi S; NABTT CNS Consortium. Immunosuppression in patients with high-grade gliomas treated with radiation and temozolomide. Clin Cancer Res. 2011 Aug 15;17(16):5473-80. doi: 10.1158/1078-0432.CCR-11-0774. Epub 2011 Jul 7. PMID 21737504
- [Result] Rudra S, Hui C, Rao YJ, Samson P, Lin AJ, Chang X, Tsien C, Fergus S, Mullen D, Yang D, Thotala D, Hallahan D, Campian JL, Huang J. Effect of Radiation Treatment Volume Reduction on Lymphopenia in Patients Receiving Chemoradiotherapy for Glioblastoma. Int J Radiat Oncol Biol Phys. 2018 May 1;101(1):217-225. doi: 10.1016/j.ijrobp.2018.01.069. Epub 2018 Feb 1. PMID 29502931
- [Result] Yovino S, Kleinberg L, Grossman SA, Narayanan M, Ford E. The etiology of treatment-related lymphopenia in patients with malignant gliomas: modeling radiation dose to circulating lymphocytes explains clinical observations and suggests methods of modifying the impact of radiation on immune cells. Cancer Invest. 2013 Feb;31(2):140-4. doi: 10.3109/07357907.2012.762780. PMID 23362951
- [Result] Paulsson AK, McMullen KP, Peiffer AM, Hinson WH, Kearns WT, Johnson AJ, Lesser GJ, Ellis TL, Tatter SB, Debinski W, Shaw EG, Chan MD. Limited margins using modern radiotherapy techniques does not increase marginal failure rate of glioblastoma. Am J Clin Oncol. 2014 Apr;37(2):177-81. doi: 10.1097/COC.0b013e318271ae03. PMID 23211224
- [Result] Minniti G, Tini P, Giraffa M, Capone L, Raza G, Russo I, Cinelli E, Gentile P, Bozzao A, Paolini S, Esposito V. Feasibility of clinical target volume reduction for glioblastoma treated with standard chemoradiation based on patterns of failure analysis. Radiother Oncol. 2023 Apr;181:109435. doi: 10.1016/j.radonc.2022.11.024. Epub 2022 Dec 16. PMID 36529439
- [Result] Singh R, Lehrer EJ, Wang M, Perlow HK, Zaorsky NG, Trifiletti DM, Bovi J, Navarria P, Scoccianti S, Gondi V, Brown PD, Palmer JD. Dose Escalated Radiation Therapy for Glioblastoma Multiforme: An International Systematic Review and Meta-Analysis of 22 Prospective Trials. Int J Radiat Oncol Biol Phys. 2021 Oct 1;111(2):371-384. doi: 10.1016/j.ijrobp.2021.05.001. Epub 2021 May 12. PMID 33991621
- [Result] Ling AL, Solomon IH, Landivar AM, Nakashima H, Woods JK, Santos A, Masud N, Fell G, Mo X, Yilmaz AS, Grant J, Zhang A, Bernstock JD, Torio E, Ito H, Liu J, Shono N, Nowicki MO, Triggs D, Halloran P, Piranlioglu R, Soni H, Stopa B, Bi WL, Peruzzi P, Chen E, Malinowski SW, Prabhu MC, Zeng Y, Carlisle A, Rodig SJ, Wen PY, Lee EQ, Nayak L, Chukwueke U, Gonzalez Castro LN, Dumont SD, Batchelor T, Kittelberger K, Tikhonova E, Miheecheva N, Tabakov D, Shin N, Gorbacheva A, Shumskiy A, Frenkel F, Aguilar-Cordova E, Aguilar LK, Krisky D, Wechuck J, Manzanera A, Matheny C, Tak PP, Barone F, Kovarsky D, Tirosh I, Suva ML, Wucherpfennig KW, Ligon K, Reardon DA, Chiocca EA. Clinical trial links oncolytic immunoactivation to survival in glioblastoma. Nature. 2023 Nov;623(7985):157-166. doi: 10.1038/s41586-023-06623-2. Epub 2023 Oct 18. PMID 37853118
- [Result] Jiang C, Mogilevsky C, Belal Z, Kurtz G, Alonso-Basanta M. Hypofractionation in Glioblastoma: An Overview of Palliative, Definitive, and Exploratory Uses. Cancers (Basel). 2023 Nov 29;15(23):5650. doi: 10.3390/cancers15235650. PMID 38067354
- [Result] Lhuillier C, Rudqvist NP, Elemento O, Formenti SC, Demaria S. Radiation therapy and anti-tumor immunity: exposing immunogenic mutations to the immune system. Genome Med. 2019 Jun 20;11(1):40. doi: 10.1186/s13073-019-0653-7. PMID 31221199
- [Result] Chajon E, Castelli J, Marsiglia H, De Crevoisier R. The synergistic effect of radiotherapy and immunotherapy: A promising but not simple partnership. Crit Rev Oncol Hematol. 2017 Mar;111:124-132. doi: 10.1016/j.critrevonc.2017.01.017. Epub 2017 Feb 4. PMID 28259287